CLINICAL TRIAL: NCT05992948
Title: Endosonograpic Monitoring of Injury to the Anal Sphincter After Transanal Stapled Anastomosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christopher Dawoud, Principal Investigator; MD, Medical University of Vienna
Other Study IDs: 2192/2019
Record Dates: First submitted 2023-03-27; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Transanal Stapled Anastomosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Transanal stapling device — Transanal stapling device used in low anterior- or anterior rectum resection, sigma resection, left hemicolectomy and intestinal reconstruction operations

SUMMARY:
Investigation of the sphincter muscles after low anterior or anterior rectum resection, and sigma resection operation by endoluminal ultrasound and manometrical examination.

ELIGIBILITY:
Inclusion Criteria:

Age 18 - 90 years, undergoing transanal stapled anastomosis at the Department of General Surgery, Medical University of Vienna

* Ability and willingness to understand and comply with study interventions and restrictions.
* Voluntarily signed informed consent after full explanation of the study to the participant.

Exclusion Criteria:

* Any physical or mental disorder, which could interfere with the participant's safety during the clinical trial or with the study objectives
* Inability to communicate well with the investigator due to language problems or reduced mental development
* Inability or unwillingness to give written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients requiring transanal stapled anastomosis due to various reasons will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
EAUS | 3 months postoperative
  Change in thickness of the anal sphincter muscles in mm from baseline to 3 months

SECONDARY OUTCOMES:
Endoanal manometry | 3 months postoperative
  Change in Anal pressure in mmHg from baseline to 3 months
EAUS2 | 3 months postoperative
  Change in the defect grade of anal sphincter muscles from baseline to 3 months
EAUS2-2 | 12 months postoperative
  Change in thickness of the anal sphincter muscles in mm from baseline to 12 months
EAUS2-2 | 12 months postoperative
  Change in the defect grade of anal sphincter muscles from baseline to 12 months
Endoanal manometry2 | 12 months postoperative
  Change in Anal pressure in mmHg from baseline to 12 months

OTHER OUTCOMES:
LARS Score | 3 months postoperative
  Change in LARS Score from baseline to 3 months
LARS Score2 | 12 months postoperative
  Change in LARS Score from baseline to 12 months
LARS2 | 12 months postoperative
  Change in LARS Score from baseline to 12 months
Vaizey Score | 3 months postoperative
  Change in Vaizey Score from baseline to 3 months
Vaizey Score2 | 12 months postoperative
  Change in Vaizey Score from baseline to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No